CLINICAL TRIAL: NCT03275181
Title: Effect of Androgen Deprivation Therapy on Left Ventricular Function in Prostate Cancer Patients and Survivors
Brief Title: Effect of Androgen Deprivation Therapy on Cardiovascular Function in Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Carl Ade, M.S., Ph.D., Assistant Professor, Kansas State University
Other Study IDs: Pro8861
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Echocardiography; Arterial Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Prostate cancer patient/survivor with ADT history: Prostate cancer patients or survivors who have a treatment history that includes androgen deprivation therapy. This includes 1) orchiectomy (surgical castration), 2) luteinizing hormone-releasing hormone (LHRH) agonists (also called LHRH analogs or Gonadotrophin-releasing hormone (GnRH) agonists), 3) LHRH antagonist, 4) CYP17 inhibitor, or 5) anti-androgen.
  Interventions: Diagnostic Test: Transthoracic Echocardiography; Diagnostic Test: Arterial blood pressure; Diagnostic Test: Submaximal Exercise
- Prostate cancer patient/survivor without ADT history: Prostate cancer patients or survivors who have never been treated with androgen deprivation therapy.
  Interventions: Diagnostic Test: Transthoracic Echocardiography; Diagnostic Test: Arterial blood pressure; Diagnostic Test: Submaximal Exercise
- Control: Individuals with no history of prostate caner androgen deprivation therapy. Free of known clinical cardiovascular disease
  Interventions: Diagnostic Test: Transthoracic Echocardiography; Diagnostic Test: Arterial blood pressure; Diagnostic Test: Submaximal Exercise

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiography — Non-invasive assessment of left ventricle structure and function
Diagnostic Test: Arterial blood pressure — Continuously monitored for 5-30 minutes via finger photoplethysmography
Diagnostic Test: Submaximal Exercise — Incremental exercise test to 85% predicted maximal heart rate on a recumbent cycle ergometer

SUMMARY:
The aim of this project is to determine whether androgen deprivation therapy (ADT) decreases left ventricular function in prostate cancer patients. If found successful, this may lead to improved cardiovascular health via treatment and/or lifestyle interventions in prostate cancer populations.

DETAILED DESCRIPTION:
Prostate Cancer is the second most common cancer among American men. Approximately 1 in 7 men will be diagnosed with prostate cancer during his lifetime. In prostate cancer patients alone, hypotestosteronemia, caused by prostate cancer treatment is associated with visceral adiposity, insulin resistance, metabolic syndrome, decreased high-density lipoprotein, increased low-density lipoprotein, increased triglycerides, loss of muscle mass, erectile disfunction, and a loss of microvascular endothelial function. Recently, several population-based studies have reported an association between androgen deprivation therapy and an increased risk of cardiovascular events, that include myocardial infarction and cardiovascular mortality. Given this link and the growing evidence that androgen-deprivation therapy adversely affects traditional risk factors, it is essential to better understand the role this type of treatment has on cardiac structure and function. As such, the manifestation of cardiovascular toxicities with prostate cancer treatment will initially be subclinical (left ventricular function changes in asymptomatic individuals) compared to clinical (including coronary symptoms or heart failure) and may develop subacutely (during treatment) or chronically.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* (Group 1) Diagnosed prostate cancer patient/survivor with a history of androgen deprivation therapy treatment
* (Group 2) Diagnosed prostate cancer patient/survivor with no history of androgen deprivation therapy treatment
* (Group 3) Cancer free

Exclusion Criteria:

* History of clinical cardiovascular disease (Atherosclerotic cardiovascular disease (ASCVD) defined by history of acute coronary syndromes, myocardial infarction (MI), stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemia attack (TIA), or peripheral arterial disease presumed to be of atherosclerotic origin)
* Not met the above criteria
* Unable to provide informed consent
* History of smoking (within 6 months) or current smoker
* Major signs or symptoms suggestive of cardiovascular, pulmonary, or metabolic disease. These include pain, discomfort in the chest, neck, jaw, arms or other areas that may result form ischemia; shortness of breath at rest or with mild exertion; Dizziness or syncope; Orthopnea or paroxysmal nocturnal dyspnea; ankle edema; palpitations or tachycardia; intermittent claudication; known heart murmur; unusual fatigue or shortness of breath with usual activities

Ages: 21 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (Experimental Group #1) Diagnosed prostate cancer patients/survivors who have received androgen deprivation therapy, (Experimental Group #2) Diagnosed prostate cancer patients/survivors who have not received androgen deprivation therapy, and (Experimental Group #3) an aged matched, healthy control group.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 1 day
  measure of left ventricular systolic function
Left ventricular strain rate | 1 day
  measure of left ventricular systolic and diastolic function

SECONDARY OUTCOMES:
Cardiac output | 1 day
  measure of cardiac function at rest and during submaximal exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas State University - Clinical Integrative Physiology Laboratory, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine GN, D'Amico AV, Berger P, Clark PE, Eckel RH, Keating NL, Milani RV, Sagalowsky AI, Smith MR, Zakai N; American Heart Association Council on Clinical Cardiology and Council on Epidemiology and Prevention, the American Cancer Society, and the American Urological Association. Androgen-deprivation therapy in prostate cancer and cardiovascular risk: a science advisory from the American Heart Association, American Cancer Society, and American Urological Association: endorsed by the American Society for Radiation Oncology. Circulation. 2010 Feb 16;121(6):833-40. doi: 10.1161/CIRCULATIONAHA.109.192695. Epub 2010 Feb 1. No abstract available. PMID 20124128
- [Background] Veccia A, Maines F, Kinspergher S, Galligioni E, Caffo O. Cardiovascular toxicities of systemic treatments of prostate cancer. Nat Rev Urol. 2017 Jan 24;14(4):230-243. doi: 10.1038/nrurol.2016.273. Online ahead of print. PMID 28117849
- [Background] Gilbert SE, Tew GA, Bourke L, Winter EM, Rosario DJ. Assessment of endothelial dysfunction by flow-mediated dilatation in men on long-term androgen deprivation therapy for prostate cancer. Exp Physiol. 2013 Sep;98(9):1401-10. doi: 10.1113/expphysiol.2013.073353. Epub 2013 May 10. PMID 23666791